CLINICAL TRIAL: NCT02644278
Title: An Open-Label, Phase 1, First-in-Human Study of the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of VX-984 in Combination With Chemotherapy in Subjects With Advanced Solid Tumors
Brief Title: First-in-Human Study of the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of VX-984 in Combination With Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201926-0001; VX15-984-001 (Other: Other)
Record Dates: First submitted 2015-12-10; First posted 2015-12-31 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-07

CONDITIONS: Advanced Solid Tumor
Keywords: VX15-984-001; VX-984; M9831; Advanced Solid Tumor; Pegylated liposomal doxorubicin
MeSH Terms: interventions — 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: FDA-regulated Device: No

ARMS (4):
- VX-984 120 mg + PLD 40 mg/m^2 (Experimental)
  Interventions: Drug: VX-984 120 mg + PLD 40 mg/m^2
- VX-984 240 mg + PLD 40 mg/m^2 (Experimental)
  Interventions: Drug: VX-984 240 mg + PLD 40 mg/m^2
- VX-984 480 mg + PLD 40 mg/m^2 (Experimental)
  Interventions: Drug: VX-984 480 mg + PLD 40 mg/m^2
- VX-984 720 mg + PLD 40 mg/m^2 (Experimental)
  Interventions: Drug: VX-984 720 mg + PLD 40 mg/m^2

INTERVENTIONS:
Drug: VX-984 120 mg + PLD 40 mg/m^2 — Participants received VX-984 orally 120 milligram (mg) orally once daily alone on Days -14 to -12 of a 14-day Lead-in Period, followed by VX-984 120 mg in combination with pegylated liposomal doxorubicin (PLD) 40 milligram per square meter (mg/m^2) administered intravenous infusion, with PLD administered on Day 1 and VX-984 administered on Day 2 to Day 4 for up to six 28-day cycle or until disease progression unacceptable toxicities, withdrawal of consent, or until exposure to PLD exceeded 550 mg/m^2.
  Other Names: M9831
  Arms: VX-984 120 mg + PLD 40 mg/m^2
Drug: VX-984 240 mg + PLD 40 mg/m^2 — Participants received VX-984 orally 240 mg orally once daily alone on Days -14 to -12 of a 14-day Lead-in Period, followed by VX-984 240 mg in combination with PLD 40 mg/m^2 administered intravenous infusion, with PLD administered on Day 1 and VX-984 administered on Day 2 to Day 4 for up to six 28-day cycle or until disease progression unacceptable toxicities, withdrawal of consent, or until exposure to PLD exceeded 550 mg/m^2.
  Arms: VX-984 240 mg + PLD 40 mg/m^2
Drug: VX-984 480 mg + PLD 40 mg/m^2 — Participants received VX-984 orally 480 mg orally once daily alone on Days -14 to -12 of a 14-day Lead-in Period, followed by VX-984 480 mg in combination with PLD 40 mg/m^2 administered intravenous infusion, with PLD administered on Day 1 and VX-984 administered on Day 2 to Day 4 for up to six 28-day cycle or until disease progression unacceptable toxicities, withdrawal of consent, or until exposure to PLD exceeded 550 mg/m^2.
  Arms: VX-984 480 mg + PLD 40 mg/m^2
Drug: VX-984 720 mg + PLD 40 mg/m^2 — Participants received VX-984 orally 720 mg orally once daily alone on Days -14 to -12 of a 14-day Lead-in Period, followed by VX-984 720 mg in combination with PLD 40 mg/m^2 administered intravenous infusion, with PLD administered on Day 1 and VX-984 administered on Day 2 to Day 4 for up to six 28-day cycle or until disease progression unacceptable toxicities, withdrawal of consent, or until exposure to PLD exceeded 550 mg/m^2.
  Arms: VX-984 720 mg + PLD 40 mg/m^2

SUMMARY:
The purpose of this study was to evaluate the safety and tolerability of VX-984 (M9831) administered alone and in combination with pegylated liposomal doxorubicin (PLD), and to determine the maximum tolerated dose (MTD) and preliminary evidence of efficacy of VX-984 in combination with PLD in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants (male and female for Part A and female for Part B) were at least 18 year of age.
* Part A Participants with histologically or cytologically confirmed malignant advanced solid tumors, who had progressed on at least 1 prior chemotherapy, and for whom either

  1. No standard care available
  2. PLD at the dose and schedule being used might be considered standard of care
* Part B

  1. Participants with histologically confirmed advanced primary endometrial cancer (locally advanced and incurable endometrial cancer that had been treated with surgery and/or radiation or is ineligible for such treatment), or recurrent or metastatic endometrial cancer, and
  2. Completed 1 line of chemotherapy treatment with a platinum-containing regimen in the advanced setting
* Measurable disease according to RECIST criteria (Version 1.1)
* Life expectancy of at least 12 weeks
* Hematological and biochemical indices within acceptable ranges shown at screening.
* Normal left ventricular ejection fraction on screening assessed by transthoracic echocardiogram or multiple gated acquisition (MUGA) scan

Exclusion Criteria:

* Previous radiotherapy (unless brachytherapy), endocrine therapy, chemotherapy, or exposure to investigational medicinal products during the 4 weeks (6 weeks for nitrosoureas and Mitomycin-C) or 4 drug half-lives before the planned administration of the first dose of study drug, whichever is greater. Previous immunotherapy during the 4 weeks before the planned administration of the first dose of study drug.
* For Part B only:

  1. Participants with uterine carcinosarcoma
  2. Prior anthracycline therapy
  3. More than 1 prior chemotherapy regimen (a participant was received first- line carboplatin and taxane and then received the same taxane second- line were considered to have had 1 prior chemotherapy regimen)
* Unresolved toxicity of Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or greater from previous anti-cancer therapy or radiotherapy
* History of spinal cord compression or brain metastases, unless asymptomatic, treated, stable, and not requiring treatment with steroids for at least 4 weeks before the planned administration of the first dose of study drug. Any history of leptomeningeal metastases.
* Female participants who was pregnant or lactating at Screening, or planned to become pregnant while on study or within 6 months after the last dose of study drug
* Female participants of childbearing potential were adhere to contraception guidelines as outlined in the protocol. Female participants were considered to be of nonchildbearing potential if they had undergone surgical hysterectomy or bilateral oophorectomy or had been amenorrheic for more than 2 years with a screening serum follicle-stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females
* Male participants with pregnant or lactating partners or partners who planned to become pregnant while on study or within 6 months after the planned administration of the last dose of study drug
* Major surgery ≤4 weeks before first dose of study drug, or incomplete recovery from a prior major surgical procedure
* Cardiac conditions
* Prior bone marrow transplant
* Extensive radiotherapy (to greater than 15% of bone marrow)
* Any other condition that in the investigator's opinion would not make the participant a good candidate for the clinical study,
* Part B: Current active malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Prior cancer in remission for 2 years or more would not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc., a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (5):
- United States (5):
  - Scottsdale, Arizona
  - Boston, Massachusetts
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First Participant First Visit: 29 Feb 2016-Last Participant Last Visit: 19-Oct-2017; A total of 15 participants were enrolled in Part A and no participants were enrolled for Part B as the study was discontinued during dose escalation in Part A, based on business related reasons as decided by the Sponsor.
Groups:
- VX-984 120 mg + PLD 40 mg/m^2: Participants received VX-984 orally 120 milligram (mg) once daily alone on Days -14 to -12 of a 14-day Lead-in Period, followed by VX-984 120 mg in combination with pegylated liposomal doxorubicin (PLD) 40 milligram per square meter (mg/m^2) administered intravenous infusion, with PLD administered on Day 1 and VX-984 administered on Day 2 to Day 4 for up to six 28-day cycle or until disease progression unacceptable toxicities withdrawal of consent, or until exposure to PLD exceeded 550 mg/m^2.
Period: Overall Study
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Started | 3 | 3 | 6 | 3
Completed | 3 | 3 | 6 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who had received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.0 (17.32) | 68.7 (5.77) | 57.5 (9.09) | 64.3 (8.33) | 59.8 (11.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 3 | 14
  Male | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 3 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 2 | 5 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-Emergent adverse events (TEAEs) were defined as AEs that were reported or worsened on or after the start of study drug dosing through the 28-day Safety Follow-up visit. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to 28 days after the last dose of study treatment, assessed up to 53.1 weeks
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants
  Any TEAE | 3 | 3 | 6 | 3
  Any Serious TEAE | 2 | 0 | 3 | 1

2. Primary Outcome: Part A: Number of Participants Who Experienced Dose Limiting Toxicity (DLT)
Description: DLT was defined using National cancer Institute Common Toxicity Criteria for Adverse Events Version 4.0 as any of the following toxicities: Grade 4 neutropenia for more than 7 days; Grade greater than or equal to (>=) 3 febrile neutropenia; Grade 4 or Grade 3 thrombocytopenia with bleeding. Grade >= 3 uncontrolled nausea/vomiting and/or diarrhea despite adequate and optimal treatment and Grade >= 3 any non- hematological adverse event (AE), except the aforementioned gastrointestinal events and alopecia.
Time Frame: Cycle 1 (each cycle is 28 days)
Population: DLT evaluable set included all participants in the safety analysis set who either met the minimum exposure criterion and had sufficient safety evaluations (as determined by the Investigators and the Sponsor) or have had a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 5 | 3
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Part A: Number of Participants With Toxicity Grade 3 or Higher in Laboratory Abnormalities
Description: The laboratory measurements included hematology and serum chemistry. It had been graded according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 into Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (Life-threatening) and Grade 5 = death. Participants with grade 3 or higher were reported.
Time Frame: Baseline up to 28 days after the last dose of study treatment, assessed up to 53.1 weeks
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants
  Participants With Hematology Abnormalities | 1 | 0 | 5 | 2
  Participants With Serum Chemistry Abnormalities | 1 | 1 | 2 | 1

4. Primary Outcome: Part A: Maximum Tolerated Dose (MTD) of VX-984 in Combination With Pegylated Liposomal Doxorubicin (PLD)
Description: The MTD was defined as the combination dose associated with the highest probability that Dose limiting toxicity (DLT) events will occur in 16.6 percent to less than 33.3 percent participants as the combination dose that not exceeded the overdose criterion (more than 25 percent probability that DLT events occurred less than or equal to (>=) 33 percent of participants. DLT was defined using National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.0.
Time Frame: Up to Cycle 1 Day 28 (each cycle is 28 days)
Population: as for outcome 2
Measure: Number; unit: milligram
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 5 | 3
milligram | NA — Due to premature discontinuation of the study, MTD was not determined. | NA — Due to premature discontinuation of the study, MTD was not determined. | NA — Due to premature discontinuation of the study, MTD was not determined. | NA — Due to premature discontinuation of the study, MTD was not determined.

5. Secondary Outcome: Part A: Area Under Plasma Concentration (AUC) During a Dosing Interval of VX-984
Description: AUC is the area under the plasma concentration curve within 1 dosing interval.
Time Frame: Pre-dose and at 0.5, 1, 2, 4, 8, and 24 hours post-dose on Day -12 and Day 4 in Cycle 1; Pre-dose and at 0.5, 1, 2, 4 hours post-dose on Day 2 in Cycle 1 (each Cycle is of 28 days)
Population: The Pharmacokinetic (PK) analysis included all participants who had received at least 1 dose of VX-984 or PLD and provided at least 1 measurable post dose concentration of VX-984 or one measurable post dose concentration of PLD.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
nanogram hour per milliliter (ng*h/mL) | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound.

6. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of VX-984
Description: Pharmacokinetic PK parameter Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
ng/mL | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound.

7. Secondary Outcome: Part A: Time to Reach Maximum Plasma Concentration (Tmax) of VX-984
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
hours | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound.

8. Secondary Outcome: Part A: Minimum Observed Plasma Concentration During Dosing Interval (Cmin) of VX-984
Description: Cmin is minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
ng/mL | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound.

9. Secondary Outcome: Part A: Area Under the Plasma Concentration Curve From Time Zero to 96 Hours Post Dose AUC(0-96h) of Pegylated Liposomal Doxorubicin
Description: The AUC(0-96h) was estimated by determining the total area under the curve of the concentration versus curve extrapolated from 0 to 96 hours.
Time Frame: Pre-infusion and at 1, 2, 4, 6, 24, 72 and 96 hours after infusion in Cycle 1 (each Cycle is of 28 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
ng*h/mL | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound.

10. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax0-96h) From Time Zero to 96 Hours Post Dose of Pegylated Liposomal Doxorubicin
Description: Cmax is the maximum observed plasma concentration obtained directly from concentration versus time curve from zero to 96 hours
Time Frame: Pre-infusion and at 1, 2, 4, 6, 24, 72 and 96 hours after infusion in Cycle 1 (each Cycle is of 28 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
ng/mL | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA (NA) — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound.

11. Secondary Outcome: Part A: Time to Reach Maximum Plasma Concentration From Zero to 96 Hours Post Dose (tmax0-96h) of Pegylated Liposomal Doxorubicin
Description: Tmax is time to reach maximum observed plasma concentration obtained directly from the concentration versus time curve from zero to 96 hours post dose.
Time Frame: Pre-infusion and at 1, 2, 4, 6, 24, 72 and 96 hours after infusion in Cycle 1 (each Cycle is of 28 days)
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
Hours | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound. | NA [NA to NA] — Although PK samples were collected, PK samples were not analyzed due to business reasons of no longer developing the compound.

12. Secondary Outcome: Part A: Number of Participants With Best Overall Response Evaluated by Response Criteria Evaluation (RECIST 1.1)
Description: The best overall response was defined as the number of participants who had achieved complete response (CR) or partial response (PR) as the best overall response according to radiological assessments as adjudicated by the IRC from randomization until the first occurrence of progressive disease (PD). CR: Complete Response (CR) defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started.
Time Frame: Up to 2 years
Population: Full analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 0 | 0
  Stable disease | 1 | 0 | 4 | 1
  Progressive disease | 0 | 3 | 0 | 1
  Not evaluable | 1 | 0 | 2 | 1

13. Primary Outcome: Part A: Number of Participants With Clinical Significant Abnormalities in Vital Signs
Description: Vital signs assessment included blood pressure, pulse rate and body temperature. Clinical significance was determined by the investigator. Number of participants with clinical significant abnormalities in vital Signs reported here.
Time Frame: Baseline up to 28 days after the last dose of study treatment, assessed up to 53.1 weeks
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0

14. Primary Outcome: Part A: Number of Participants With Clinical Significant Abnormalities Echocardiograms
Description: Echocardiogram is a graphic outline of the heart's movement. Clinical significance was determined by the investigator. Number of participants with clinical significant abnormalities in Echocardiograms reported here.
Time Frame: Baseline up to 28 days after the last dose of study treatment, assessed up to 53.1 weeks
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0

15. Primary Outcome: Part A: Number of Participants With Clinical Significant Abnormalities in Electrocardiogram(ECG) Parameters
Description: ECG parameters included heart rate, pulse rate, QRS,QT, RR, QTcB and QTcF. Clinical significance was determined by the investigator. Number of participants with clinical significant abnormalities in ECG parameters reported here.
Time Frame: Baseline up to 28 days after the last dose of study treatment, assessed up to 53.1 weeks
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
Number analyzed (Participants) | 3 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days of follow up after the last dose of study treatment, assessed up to 53.1 weeks
Arm/Group | VX-984 120 mg + PLD 40 mg/m^2 | VX-984 240 mg + PLD 40 mg/m^2 | VX-984 480 mg + PLD 40 mg/m^2 | VX-984 720 mg + PLD 40 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 2/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 3/6 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-984 120 mg + PLD 40 mg/m^2 (N=3) | VX-984 240 mg + PLD 40 mg/m^2 (N=3) | VX-984 480 mg + PLD 40 mg/m^2 (N=6) | VX-984 720 mg + PLD 40 mg/m^2 (N=3)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-984 120 mg + PLD 40 mg/m^2 (N=3) | VX-984 240 mg + PLD 40 mg/m^2 (N=3) | VX-984 480 mg + PLD 40 mg/m^2 (N=6) | VX-984 720 mg + PLD 40 mg/m^2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 4 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 2
Asthenia (General disorders) | 0 | 1 | 2 | 0
Fatigue (General disorders) | 2 | 2 | 2 | 3
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 1 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 2 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was discontinued during dose escalation in Part A, based on business related reasons as decided by the Sponsor. Therefore, the expansion cohorts (Part B) were not conducted. Hence, we have not reported the outcome measure of Part B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT02644278/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/78/NCT02644278/SAP_001.pdf